CLINICAL TRIAL: NCT01878149
Title: Retrospective Multicenter Clinical Evaluation of Complications for Single or Multilevel VEO® Lateral Access and Interbody Fusion System and eXtreme Lateral Interbody Fusion (XLIF®) Subjects
Status: Completed | Type: Observational
Sponsor: Baxano Surgical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PR-0025; PR-0025 (Other: TranS1)
Record Dates: First submitted 2013-06-11; First posted 2013-06-14 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VEO® Lateral Access and Interbody Fusion System
- eXtreme Lumbar Interbody Fusion (XLIF®)

SUMMARY:
The purpose of this retrospective clinical evaluation is to compare VEO® single or multilevel results to XLIF® single or multilevel results relative to the safety endpoints. This study will collect retrospective data on subjects who were treated with VEO® and XLIF® at least 3 months prior to the initiation of this study. Given that fusion generally takes at least 6 months to determine, the aim of this study is not to determine fusion but to consider the short-term (out to 6 months) reported adverse events between the two cohorts.

Devices used in both systems are cleared for use and conform to US regulatory requirements. The study employs these procedures and devices for uses that are consistent with their 510(k), legally cleared, labeling.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older;
* Male or female VEO® subjects that had previously received the single or two level LLIF procedure using the VEO® or XLIF® systems as an adjunct to fusion at L2-S1 to treat degenerative disc disease (DDD) at the treated level;
* Subject that was treated no less than 3 months prior to this evaluation with the LLIF procedure using the VEO® or XLIF® system by the participating surgeons.

Exclusion Criteria:

* Subject who did not receive LLIF procedure using the VEO® or XLIF® system for fusion of L2-S1;
* Subjects with less than 3 months of follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 40 subjects will be enrolled across the participating sites; 20 subjects who have been treated with the VEO® lateral system and 20 who have been treated with the XLIF® system. Consecutive subjects at the participating sites that meet all of the inclusion criteria and none of the exclusion criteria will be eligible for study participation until the enrollment target is reached.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Yuan, MD, Principal Investigator — Memorial Orthopaedic Surgical Group
Locations (4):
- United States (4):
  - Memorial Orthopaedic Surgical Group, Long Beach, California
  - Minimally Invasive Neurosurgery, Santa Ana, California
  - NorthShore LIJ, Great Neck, New York
  - Advanced Spine & Pain, Arlington, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consecutive subjects at each site meeting all of the study eligibility criteria and who were treated with LLIF using the VEO® or XLIF® systems at least 3 months prior to the date the data is collected were included in this evaluation.
Pre-assignment Details: The Sponsor originally collected data on 38 subjects, 21 subjects in the VEO treatment arm and 17 subjects in the XLIF® treatment arm, from a total of five sites. Four study subjects (two subjects from each study arm) were excluded from the final evaluation as they did not meet the inclusion/exclusion criteria.
Groups:
- VEO® Lateral Access and Interbody Fusion System: VEO® is the brand name for the Baxano Surgical LLIF system, which employs traditional LLIF patient positioning, disc space preparation, implant placement, and is compatible with neuromonitoring. The VEO® system was developed with an initial, radiolucent retractor that is placed at the psoas fascia and held in place with an articulated arm. Dissection through the psoas is then performed with direct vision in conjunction with EMG. The psoas muscle is split anterior-posterior along muscle fiber lines and the retraction is performed with two independent blades. Insertion depth may be varied to avoid muscle creep, and the toed-out blade tips are positioned under the psoas to hold the system in place. An inner sleeve is inserted to lock the blades in place at the desired radial tension for a customizable disc space exposure. Standard discectomy, endplate preparation, cage implantation, and wound closure are performed.
- eXtreme Lumbar Interbody Fusion (XLIF®): The eXtreme lumbar interbody fusion (XLIF®) is the brand name of the LLIF system distributed by NuVasive®, Inc.When the XLIF® system is used for LLIF, the patient is placed in the lateral decubitus position and the retroperitoneal space is accessed through blunt dissection. Using proprietary neuromonitoring, a series of graduated muscle dilators are advanced through the psoas muscle down to the disc space at the lumbar level of interest. Real-time EMG evoked potential values indicate proximity of motor nerves to direct safe dilator placement. A guidewire is placed into the disc space through the initial cannulated dilator to fix retractor placement. A psoas muscle retractor system is inserted over the dilators and blades are carefully opened over the disc space in the caudal-cephalad and anterior directions under direct live EMG. Upon achieving sufficient disc space exposure, standard discectomy, endplate preparation, cage implantation, and wound closure are performed.
Period: Overall Study
Arm/Group | VEO® Lateral Access and Interbody Fusion System | eXtreme Lumbar Interbody Fusion (XLIF®)
Started | 21 | 17
Completed | 19 | 15
Not Completed | 2 | 2
Not completed — Did Not Meet Eligibility Criteria | 2 | 2

BASELINE CHARACTERISTICS:
Population: Given the nature of this retrospective evaluation, the sample size was not statistically derived but was instead intended to be representative of the body of evidence that exist for real world usage of the VEO® device.
Groups:
- VEO® Lateral Access and Interbody Fusion System: This study included adult men and women (> 18 years old) who received a lateral lumbar interbody fusion (LLIF) with the VEO® spinal procedure. VEO® is intended to treat patients with conditions who typically require fusion at the lumbar levels for degenerative disc disease (DDD).
- eXtreme Lumbar Interbody Fusion (XLIF®): This study included adult men and women (> 18 years old) who received a lateral lumbar interbody fusion (LLIF) with the XLIF® spinal procedure. XLIF® is intended to treat patients with conditions who typically require fusion at the lumbar levels for degenerative disc disease (DDD).
- Total: Total of all reporting groups
Arm/Group | VEO® Lateral Access and Interbody Fusion System | eXtreme Lumbar Interbody Fusion (XLIF®) | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.63 (13.13) | 63 (12.35) | 62.21 (12.36)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 17
  Male | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  United States | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants Without Major Device-related Adverse Events and/or Failures
Description: Incidence of major device-related adverse events and/or failures, defined as those requiring revision surgery or a secondary operation, or events resulting in permanent disability or death.
Time Frame: Observed for up to 6 months post-surgery
Population: It was anticipated that approximately 40 subjects would be enrolled across the participating sites; 20 subjects in each treatment arm. Consecutive subjects who were treated with LLIF using the VEO® or XLIF® systems at least 3 months prior to the the data collection were included. The planned sample size was not statistically derived.
Measure: Number; unit: participants
Groups:
- VEO® Lateral Access and Interbody Fusion System: VEO® is the brand name for the LLIF system introduced by Baxano Surgical® in 2011. The VEO Lateral system employs traditional LLIF patient positioning, disc space preparation, implant placement, and is compatible with neuromonitoring. However, the VEO® system posesses a radiolucent retractor that is placed at the psoas fascia and held in place with an articulated arm. This retractor was developed to address the reliance on EMG neuromonitoring alone with traditional LLIF approaches to avoid injury to lumbar plexus nerve roots, particularly as EMG is limited to monitoring motor nerves. Moreover, there was a desire to avoid reliance on fluoroscopy alone to determine retractor placement, without significant assessment of intervening anatomy.
- eXtreme Lumbar Interbody Fusion (XLIF®): The eXtreme lumbar interbody fusion (XLIF®) is the brand name of the LLIF system distributed by NuVasive®, Inc. in 2001. When the XLIF® system is used for LLIF, the patient is placed in the lateral decubitus position and the retroperitoneal space is accessed through blunt dissection. Using proprietary neuromonitoring, a series of graduated muscle dilators are advanced through the psoas muscle down to the disc space at the lumbar level of interest. Real-time EMG evoked potential values indicate proximity of motor nerves to direct safe dilator placement. A guidewire is placed into the disc space through the initial cannulated dilator to fix retractor placement. A psoas muscle retractor system is inserted over the dilators and the blades are carefully opened over the disc space in the caudal-cephalad and anterior directions under direct live EMG. Upon achieving sufficient disc space exposure, standard discectomy, endplate preparation, cage implantation, and wound closure are performed.
Arm/Group | VEO® Lateral Access and Interbody Fusion System | eXtreme Lumbar Interbody Fusion (XLIF®)
Number analyzed (Participants) | 19 | 15
participants | 19 | 15

2. Secondary Outcome: Safety
Description: Incidence of short term peri-operative adverse events (out to 6 months post-implant) including thigh pain, numbness, paresthesia and transient leg weakness.
Time Frame: Observed for up to 6 months post-surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- VEO® Lateral Access and Interbody Fusion System: VEO® is the brand name for the LLIF system introduced by Baxano Surgical® in 2011. The VEO® Lateral system employs traditional LLIF patient positioning, disc space preparation, implant placement, and is compatible with neuromonitoring. However, the VEO® system posesses a radiolucent retractor that is placed at the psoas fascia and held in place with an articulated arm. This retractor was developed to address the reliance on EMG neuromonitoring alone with traditional LLIF approaches to avoid injury to lumbar plexus nerve roots, particularly as EMG is limited to monitoring motor nerves. Moreover, there was a desire to avoid reliance on fluoroscopy alone to determine retractor placement, without significant assessment of intervening anatomy.
Arm/Group | VEO® Lateral Access and Interbody Fusion System | eXtreme Lumbar Interbody Fusion (XLIF®)
Serious Adverse Events (participants affected / at risk) | 0/21 | 4/17
Other Adverse Events (participants affected / at risk) | 8/21 | 7/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VEO® Lateral Access and Interbody Fusion System (N=21) | eXtreme Lumbar Interbody Fusion (XLIF®) (N=17)
Deep venous thrombosis and GI prophylaxis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Renal vein nicked (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Respiratory failure on a ventilator (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Severe Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Severe blood loss of 1000 mL
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VEO® Lateral Access and Interbody Fusion System (N=21) | eXtreme Lumbar Interbody Fusion (XLIF®) (N=17)
Lower extremity weakness (Nervous system disorders) | 3 (3) | 1 (1) — Lower extremity weakness
Decreased strength (Nervous system disorders) | 0 (0) | 1 (1) — Decreased Strength
Lower extremity numbness (Nervous system disorders) | 5 (5) | 3 (3) — Lower extremity numbness
Lower extremity pain (Nervous system disorders) | 3 (3) | 4 (4) — Lower extremity pain includes pain of the leg, thigh, hip, buttocks, and groin
Parasthesia (Nervous system disorders) | 0 (0) | 1 (1) — Parasthesia
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Incisional Pain (Surgical and medical procedures) | 0 (0) | 1 (1)
Wound infection (Surgical and medical procedures) | 0 (0) | 2 (2)
Limited flexion/extension at waist (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Severe bleeding (Surgical and medical procedures) | 0 (0) | 1 (1) — Severe blood loss of 1000 mL during surgery
Renal vein nicked (Surgical and medical procedures) | 0 (0) | 1 (1) — Renal vein nicked during surgery
Wound ecchymosis (Surgical and medical procedures) | 0 (0) | 1 (1) — Minimal ecchymosis around wound
Respiratory failure (Surgical and medical procedures) | 0 (0) | 1 (1) — Respiratory failure on ventilator
Deep venous thrombosis prophylaxis and GI prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less